CLINICAL TRIAL: NCT04316052
Title: Comparing the Effect of Aerobic And Strength Training Exercises For Restless Leg Syndrome In Patients With Diabetes
Brief Title: Aerobic And Strength Training Exercises For Restless Leg Syndrome In Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00660 Fizah Mahnoor
Record Dates: First submitted 2020-03-06; First posted 2020-03-20 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Restless Legs Syndrome; Diabetes
Keywords: RLS,; Diabetes,; Aerobic training,; strength training
MeSH Terms: conditions — Restless Legs Syndrome; Diabetes Mellitus | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic training group (Experimental): At the visit, participants will be first instructed in the use of the treadmill, which included heart rate assessment capability. Walking intensity and duration prescriptions will be accordance with recommendations of the American College of Sports Medicine.
  Interventions: Other: Aerobic training
- strength training group (Experimental): Strength training prescriptions will be in accordance with recommendations of the American College of Sports Medicine.
  Interventions: Other: strength training

INTERVENTIONS:
Other: Aerobic training — After the baseline assessment, Following randomization into the exercise group, participants will undergo an exercise program orientation, which will be conducted individually.At the visit, participants will be first instructed in the use of the treadmill, which included heart rate assessment capability. Walking intensity and duration prescriptions will be accordance with recommendations of the American College of Sports Medicine. Participants will be instructed to walk for 45 minutes, including a 5-minute warm-up and 5 min cool-down, at 50% to 80% of their age-predicted maximum heart rate.Over the course of 4 months, each patient will complete 48 sessions. The morning after the 24th and 48nd sessions of aerobic physical exercise, each participant will be assessed completely
  Arms: aerobic training group
Other: strength training — After the baseline assessment, participants will undergo exercise program orientation, which will be conducted individually. Participants will be instructed to perform 45 min session, two sets of 8 to 12 repetitions of each exercise (2 second hold each up and down hold) for the first 2 weeks to provide an introductory period. In the first session, muscular strength will be assessed using a standardized 10-repetition maximum approach, from which one repetition maximum (1-RM) will be estimated. The exercise prescription for strength training will be made at approximately 50% of the estimated 1-RM.The strength training activities included horizontal leg press, leg extension, leg curl, hip adduction, hip abduction, and seated rotary calf press.
  Arms: strength training group

SUMMARY:
The aim of this research is to find and compare the effect of aerobic exercises and strength training exercise on RLS severity in diabetic patient. Randomized controlled trials done at Physical therapy department of Pakistan Railway general hospital, Rawalpindi. The sample size was 38.The subjects were divided into two groups, 19 subjects in the aerobic physical therapy group and in 19 strength group. Study duration was of 6 months. Sampling technique applied was Simple randomization via computer-generated random numbers. Only 40-60 years individual with restless leg syndrome in 5 years old diabetic history included. Tools used in the study are International Restless Leg Syndrome Study Group Rating Scale: (an International tool for finding the severity of RLS), The Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESS). Data was be analyzed through SPSS 21.

DETAILED DESCRIPTION:
Restless legs syndrome (RLS) is a common, underdiagnosed neurological movement disorder of undetermined aetiology. RLS is a collective sensory-motor neural condition that is described by deep restlessness, unpleasant creeping/crawling perceptions profound inside the lower limbs and sleep disturbance, accompanied by a need to move the limb often at bedtime. Usually, the sensory-motor complaints of Restless Leg Syndrome arise or aggravate nocturnally, presenting a day-to-day pattern. These sensations typically occur before sleep onset and cause sleep disturbance in patients. Restless leg syndrome is associated with different conditions including diabetes, diabetic neuropathy, pregnancy, uremia, iron deficiency, hypertension and coronary heart diseases. The Pathophysiology of restless leg syndrome is not clear. Firstly, it was thought to be peripheral nerve disorder, later in last two eras, the authors agreed that origin of Restless Leg Syndrome is in Central Nervous System and there is variation in complex combination between CNS and PNS structures. There is an unusual sensory-motor combination and boosted spinal cord impulsiveness. The positive outcomes of the dopaminergic treatment show that restless leg syndrome may be caused by dopamine dysfunction and iron deficiency in CNS. Prevalence of RLS was found 27%.

One of the most important risk factors of RLS is diabetes. According to a study by in 2019 stated Diabetes type 2 prevalence is 80.0%. Various Studies on Restless Leg Syndrome in diabetes is conducted showing a significant association between RLS and type 2 diabetes. A study was done in Saudi Arabia reported that RLS can affect diabetic patients and it is important to treat RLS, for even better diabetes control. Prevalence of RLS in diabetic patient is 28.6%. Mostly RLS is mixed with other sleep disorder known as a periodic limb movement disorder. Restless leg syndrome also causes strong sleep disturbances (e.g., chronic insomnia, sleep apnea) which have a major impact on health and quality of life, its adverse impact can usually be reversed by on-time diagnosis and treatment. The primary treatments for restless legs syndrome are pharmacological but recently non-pharmacological treatment is being used. A single-blinded RCT was done in 2013 on the physical therapy management of restless leg syndrome in hemodialysis patients stated progressive exercise training program appears to be a safe and effective approach in reducing RLS symptom severity in HD patients. It seems that exercise-induced adaptations to the whole body are mostly responsible for the reduction in RLS severity score. Another study in 2016 was done in which it was reported that muscle stretching exercise seems to be very effective and can reduce RLS symptoms. A 12-week trial in restless leg syndrome patient. The exercise group was prescribed a conditioning program of the aerobic and control group was prescribed lower-body resistance training, both groups had a positive effect on decreasing severity but the exercise group had a significant improvement in symptoms compared with the control group. Diabetes is one of the most prevalent risk factors of "Restless leg syndrome" but unluckily there were limited studies done here in Pakistan for severity control. Our study differs from other literature in sense of its an RCT investigator is trying to find out better treatment option by comparing two treatments (aerobic training and strengthening exercise) for diabetic patients suffering from restless leg syndrome.

ELIGIBILITY:
Inclusion Criteria:

* The RLS will be diagnosed using the four criteria defined by the International Restless Legs Syndrome Study Group.
* Patient with 5 years old diabetes type II history
* Both genders
* Patients with age limit 40-60 years
* Lower limb MMT 4/5

Exclusion Criteria:

* Severe Co-morbidities like Cardiac Failure, Stroke etc.
* Impaired Cognition
* Communication problems
* Infectious disease, fracture etc.
* Serious visual or hearing impairments

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
International Restless Leg Syndrome Study Group Rating Scale: (International tool for finding the severity of RLS) | 12 weeks
  This validated 10-item questionnaire was designed to assess symptom severity, frequency, and impact on daily life. RLS symptom severity score will be determined by summing the questionnaire answers. The maximum score is 40, and a higher score indicates more severe RLS. The total score on the RLS Rating Scale questionnaire will be used as the primary outcome measure of RLS severity. Validity of this scale is 0.84. Internal consistency Cronbach alpha measures is 0.93, Inter-examiner reliability is 0.95 and Test-retest reliability is 0.87. Changes will be assessed from baseline

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI). | 12 weeks
  Sleep quality can be evaluated by the Pittsburgh Sleep Quality Index (PSQI). This scale has seven components, each one dealing with a major aspect of sleep: 1) subjective quality of sleep, 2) sleep onset latency, 3) sleep duration, 4) sleep efficiency, 5) the presence of sleep disturbances, 6) the use of hypnotic or sedative medication, and 7) the presence of daytime disturbances, as an indication of daytime alertness. Individuals with a PSQI score of six or more are considered poor sleepers. The PSQI global score correlation coefficient for test - retest reliability is.87. Validity analyses showed high correlations between PSQI and sleep log data. A PSQI global score > 5 resulted in a sensitivity of 91.55.Changes will be assessed from baseline

OTHER OUTCOMES:
Epworth Sleepiness Scale (ESS) | 12 weeks
  The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness. The ESS is a self-administered questionnaire with 8 questions. The ESS asks the respondent to rate on a 4-point scale (0-3) their usual chances of having dozed off or fallen asleep while engaged in eight different activities that differ widely. The ESS score is highly correlated (r = 0.82) and the internal consistency as measured by Cronbach's alpha is 0.88. Changes will be assessed from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Aruba Saeed, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sevim S, Dogu O, Kaleagasi H, Aral M, Metin O, Camdeviren H. Correlation of anxiety and depression symptoms in patients with restless legs syndrome: a population based survey. J Neurol Neurosurg Psychiatry. 2004 Feb;75(2):226-30. PMID 14742594
- [Background] Berger K, Luedemann J, Trenkwalder C, John U, Kessler C. Sex and the risk of restless legs syndrome in the general population. Arch Intern Med. 2004 Jan 26;164(2):196-202. doi: 10.1001/archinte.164.2.196. PMID 14744844
- [Background] Nichols DA, Allen RP, Grauke JH, Brown JB, Rice ML, Hyde PR, Dement WC, Kushida CA. Restless legs syndrome symptoms in primary care: a prevalence study. Arch Intern Med. 2003 Oct 27;163(19):2323-9. doi: 10.1001/archinte.163.19.2323. PMID 14581252
- [Background] Restless legs syndrome: detection and management in primary care. National Heart, Lung, and Blood Institute Working Group on Restless Legs Syndrome. Am Fam Physician. 2000 Jul 1;62(1):108-14. PMID 10905782
- [Background] Hening W, Walters AS, Allen RP, Montplaisir J, Myers A, Ferini-Strambi L. Impact, diagnosis and treatment of restless legs syndrome (RLS) in a primary care population: the REST (RLS epidemiology, symptoms, and treatment) primary care study. Sleep Med. 2004 May;5(3):237-46. doi: 10.1016/j.sleep.2004.03.006. PMID 15165529
- [Background] Walters AS. Toward a better definition of the restless legs syndrome. The International Restless Legs Syndrome Study Group. Mov Disord. 1995 Sep;10(5):634-42. doi: 10.1002/mds.870100517. PMID 8552117
- [Background] De Mello MT, Esteves AM, Tufik S. Comparison between dopaminergic agents and physical exercise as treatment for periodic limb movements in patients with spinal cord injury. Spinal Cord. 2004 Apr;42(4):218-21. doi: 10.1038/sj.sc.3101575. PMID 15060518
- [Background] Abetz L, Allen R, Follet A, Washburn T, Earley C, Kirsch J, Knight H. Evaluating the quality of life of patients with restless legs syndrome. Clin Ther. 2004 Jun;26(6):925-35. doi: 10.1016/s0149-2918(04)90136-1. PMID 15262463
- [Background] Lopes LA, Lins Cde M, Adeodato VG, Quental DP, de Bruin PF, Montenegro RM Jr, de Bruin VM. Restless legs syndrome and quality of sleep in type 2 diabetes. Diabetes Care. 2005 Nov;28(11):2633-6. doi: 10.2337/diacare.28.11.2633. PMID 16249531
- [Background] Omar SM, Musa IR, ElSouli A, Adam I. Prevalence, risk factors, and glycaemic control of type 2 diabetes mellitus in eastern Sudan: a community-based study. Ther Adv Endocrinol Metab. 2019 Jun 27;10:2042018819860071. doi: 10.1177/2042018819860071. eCollection 2019. PMID 31275546
- [Background] Merlino G, Fratticci L, Valente M, Del Giudice A, Noacco C, Dolso P, Cancelli I, Scalise A, Gigli GL. Association of restless legs syndrome in type 2 diabetes: a case-control study. Sleep. 2007 Jul;30(7):866-71. doi: 10.1093/sleep/30.7.866. PMID 17682657
- [Background] Zobeiri M, Shokoohi A. Restless leg syndrome in diabetics compared with normal controls. Sleep Disord. 2014;2014:871751. doi: 10.1155/2014/871751. Epub 2014 May 7. PMID 24895540